CLINICAL TRIAL: NCT04076488
Title: Feasibility of an Interactive Tablet-based Exercise Program for People With Chronical Diseases
Acronym: TABEX-CD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zemp Damiano (Other)
Collaborators: Ente Ospedaliero Cantonale, Bellinzona (Other); ETH Zurich (Other)
Responsible Party: Sponsor-Investigator, Zemp Damiano, Principal Investigator, Ente Ospedaliero Cantonale, Bellinzona
Organization: Ente Ospedaliero Cantonale, Bellinzona (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2019-01161 CE 3497
Record Dates: First submitted 2019-08-16; First posted 2019-09-03 (Actual); Last update posted 2021-01-22 (Actual); Status verified 2021-01

CONDITIONS: End Stage Renal Disease
Keywords: Telemedicine; Exercise; Feasibility
MeSH Terms: conditions — Kidney Failure, Chronic; Motor Activity

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dividat FIT: Computer based exercise (Experimental): Tablet based interactive physical training.
  Interventions: Other: Dividat Fit

INTERVENTIONS:
Other: Dividat Fit — tablet based, remote assisted home-training

SUMMARY:
End Stage Renal Disease (ESRD) is a potential outcome of Chronic Kidney Disease (CKD) that requires renal replacement therapy in the form of dialysis or transplantation.Despite the encouraging benefits seen in PHD who exercised, they may be confronted with more barriers to start and maintain an exercise program than healthy persons, e.g. due to reduced accessibility of specialised physiotherapists. Telerehabilitation (TR), a subfield of telemedicine, may help to overcome some of the barriers to exercise regularly and connect PHD with specialised physiotherapists. The primary objective of this study is to determine feasibility of this TR exercise approach in preparation of a future RCT. Focus of the study is recruitment, attrition and adherence to the intervention, data collection methods and acceptability/satisfaction of the intervention.

The secondary objectives are to evaluate potential impacts of this intervention approach on physical function and health-related disability and quality of life. The study intervention is an interactive tablet-based home exercise program. The program is called "Dividat Fit" and works interactive, meaning that the responsible specialised Physiotherapist (PT) supervises the training progression of her/his patient weekly and if necessary assists the patient via remote or through a visit at home.

DETAILED DESCRIPTION:
End Stage Renal Disease (ESRD) is a potential outcome of Chronic Kidney Disease (CKD) that requires renal replacement therapy in the form of dialysis or transplantation. The prevalence rate of people undergoing dialysis is 296 of 1 Million. 90% of them receiving haemodialysis (HD). For haemodialytic therapy, patients need to receive dialyses 2-3 times a week in an outpatient hospital facility or a clinic lifelong or until kidney transplantation. A dialyses session last between 3 and 4 hours.

Nowadays, the beneficial effects of exercise in people undergoing haemodialysis (PHD) are well accepted and there is evidence that they profit from an exercise program.

Despite the encouraging benefits seen in PHD who exercised, they may be confronted with more barriers to start and maintain an exercise program than healthy persons, e.g. due to reduced accessibility of specialised physiotherapists. Telerehabilitation (TR), a subfield of telemedicine, may help to overcome some of the barriers to exercise regularly and connect PHD with specialised physiotherapists. TR is defined as the provision of rehabilitation services from a distance using telecommunication technologies as the delivery medium. This approach may optimize the timing, intensity and sequencing of interventions and provide opportunities for individuals to receive rehabilitation in their own social and professional environments from disease-specialised caregivers. An additional advantage of TR is the possibility to implement different persuasive technologies such as personalisation, self-monitoring, tailoring, goal setting, comparison and conditioning through positive and negative reinforcement in the development of exercise programmes. These technologies help to make exercise programmes more enjoyable and, therefore, enhance patients' motivation to exercise regularly.

Furthermore, the importance of individual and social support has been emphasized in several reviews evaluating health behaviour change for example becoming more active. This kind of support can be integrated in the design of a TR program.

To the best of our knowledge, there exist no TR programme especially designed for PHD. Therefore, the aim of this study is to evaluate feasibility of a tablet-based exercise program, called "Dividat Fit" for PHD.

The study intervention is an interactive tablet-based home exercise program. The program is called "Dividat Fit" and works interactive, meaning that the responsible specialised Physiotherapist (PT) supervises the training progression of her/his patient weekly and if necessary assists the patient via remote or through a visit at home.

During the first face-to-face session, the PT examines the patient, sets up an individually tailored physical exercise (PE) program with four to six exercises and practises these exercises with the patient. Before the patient will start with the 12-week home program, she/he receives a tablet-computer on which the physical exercises are programmed as well as an instruction how to use "Dividat Fit". During the whole training program, the PT tele-monitors each patient by checking the training diary weekly and providing written feedback to the exercises and the comments, if applicable. If needed, the PT contacts the participants (per phone).

10-15 participants will be recruited. For feasibility studies, a sample size calculation is not possible. There are different rules of thumb for the sample size of feasibility studies. One general rule of thumbs recommends 12 participants for a feasibility study. Another recommendation is based on the estimated effect size: they recommend 15 or 10 patients for standardized effect sizes that are medium (0.5) or large (0.8), respectively.

ELIGIBILITY:
Inclusion Criteria:

* haemodialysis patients older than 60 years
* able to walk 20 meters independently without walking aids
* currently exercising less than one training session per week
* maintenance of a stable medical regimen for 4 weeks prior to initiation of study and considered to maintain a stable regimen for the course of the study
* signed informed consent to participate in the study

Exclusion Criteria:

* clinically significant concomitant disease states
* contraindications to physical exercise
* known or suspected non-compliance, drug or alcohol abuse
* inability to follow the procedures of the study, e.g. due to language problems, psychological disorders, dementia, etc. of the participant
* participation in another study with investigational drug within the 30 days preceding and during the present study

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2020-10-29 (Actual); Study Completion 2020-10-29 (Actual)

PRIMARY OUTCOMES:
Adherence | Will be assessed approximately 6 months after start of study
  Attrition and adherence rate (attrition rate and reasons of drop-out, adherence rate, adherence to the described exercises)
Feasibility of the training | Will be assessed approximately 6 months after start of study
  Technology Acceptance Model

SECONDARY OUTCOMES:
Functional Test | At baseline and after 3 months of training
  Short Physical Performance Battery
Performance Test | At baseline and after 3 months of training
  Timed Up & Go Test

OTHER OUTCOMES:
Autonomy evaluation | At baseline and after 3 months of training
  De Morton Mobiity Index
Health and quality of life parameters | At baseline and after 3 months of training
  SF-12
Endurance | At baseline and after 3 months of training
  1 minute stand up test

CONTACTS AND LOCATIONS:
Overall Officials: Damiano Zemp, MSc, Principal Investigator — Ente Ospedaliero Cantonale, Bellinzona
Locations (1):
- Ente Ospedaliero Cantonale, Bellinzona, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zemp DD, Baschung Pfister P, Knols RH, Quadri P, Bianchi G, Giunzioni D, Lavorato S, Giannini O, de Bruin ED. A blended e-health intervention for improving functional capacity in elderly patients on haemodialysis: A feasibility study. Front Digit Health. 2022 Dec 6;4:1054932. doi: 10.3389/fdgth.2022.1054932. eCollection 2022. PMID 36561924